CLINICAL TRIAL: NCT01528735
Title: An Open-label, Ascending Dose, Phase II Study to Evaluate Tolerability, Safety, Antiviral Activity, and Pharmacokinetics of BI 207127 NA in Combination With BI 201335 NA and Ribavirin for 8 Weeks in Treatment-naïve Japanese Patients With Genotype 1chronic Hepatitis C Virus Infection
Brief Title: This Trial Evaluates Safety, Pharmacokinetic Profile and Anti-viral Response of BI 207127 and BI 201335 for Patients With Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.25
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin

ARMS (2):
- BI 207127 NA, BI 201335 NA(high dose), R (Experimental): Patients receive BI 207127 NA,BI 201335 NA(high dose) and RBV for 8 wks followed by BI 201335 NA,PegIFN/RBV for 24 wks
  Interventions: Drug: peginterferon; Drug: Ribavirin; Drug: BI 207127 NA; Drug: BI 201335 NA
- BI 207127 NA,BI 201335 NA(low dose),RBV (Experimental): Patients receive BI 207127 NA,BI 201335 NA(low dose) and RBV for 8 wks followed by BI 201335 NA,PegIFN/RBV for 24 wks
  Interventions: Drug: BI 207127 NA; Drug: Ribavirin; Drug: BI 201335 NA; Drug: peginterferon

INTERVENTIONS:
Drug: BI 207127 NA — one fix dose
  Arms: BI 207127 NA,BI 201335 NA(low dose),RBV
Drug: peginterferon — per package insert
  Arms: BI 207127 NA, BI 201335 NA(high dose), R
Drug: Ribavirin — per weight BID
  Arms: BI 207127 NA,BI 201335 NA(low dose),RBV
Drug: Ribavirin — per weight BID
  Arms: BI 207127 NA, BI 201335 NA(high dose), R
Drug: BI 207127 NA — one fix dose
  Arms: BI 207127 NA, BI 201335 NA(high dose), R
Drug: BI 201335 NA — high dose
  Arms: BI 207127 NA, BI 201335 NA(high dose), R
Drug: BI 201335 NA — low dose
  Arms: BI 207127 NA,BI 201335 NA(low dose),RBV
Drug: peginterferon — per package insert
  Arms: BI 207127 NA,BI 201335 NA(low dose),RBV

SUMMARY:
The objective of this trial is to investigate tolerability, safety, pharmacokinetics and antiviral activity of BI 207127 NA in combination with BI 201335 NA and ribavirin for 8 weeks in Japanese treatment-naive patients with chronic GT-1 HCV infection.

ELIGIBILITY:
Inclusion criteria:

* Chronic hepatitis C, diagnosed by positive anti-hepatitis C virus(HCV) antibodies and detected HCV ribonucleic acid(RNA) at screening in addition to:

  1. positive anti-HCV antibodies or detected HCV RNA at least 6 months prior to screening; or,
  2. liver biopsy consistent with chronic HCV infection.
* HCV infection of genotype 1 confirmed by genotypic testing at screening
* Therapy-naïve to interferon, pegylated interferon, ribavirin or any antiviral / immunomodulatory drug for acute or chronic HCV infection.
* Plasma HCV RNA = 100,000 IU/mL at screening

Exclusion criteria:

* Hepatitis C infection of mixed genotype (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening
* Human immunodeficiency virus (HIV) co-infection
* Decompensated liver disease, or history of decompensated liver disease
* Body weight < 40 or > 125 kg at screening
* Hemoglobin <12.0g/dL for women and <13.0g/dL for men at screening
* White blood cell count <3000 cells/mm3 at screening
* Absolute neutrophil count < 1,500 cells/mm3 at screening
* Platelet count < 90,000 /mm3 at screening
* Serum creatinine > 1.5xUpper Limit of Normal range(ULN) or creatinine clearance =50 mL/min at screening

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- Japan (5):
  - 1241.25.002 Boehringer Ingelheim Investigational Site, Kofu, Yamanashi
  - 1241.25.005 Boehringer Ingelheim Investigational Site, Kurashiki, Okayama
  - 1241.25.003 Boehringer Ingelheim Investigational Site, Nagoya, Aichi
  - 1241.25.004 Boehringer Ingelheim Investigational Site, Nishinomiya, Hyogo
  - 1241.25.001 Boehringer Ingelheim Investigational Site, Omura, Nagasaki

REFERENCES:
- [Derived] Yatsuhashi H, Kodani N, Ugai H, Omata M. Open-label phase 2 study of faldaprevir, deleobuvir and ribavirin in Japanese treatment-naive patients with chronic hepatitis C virus genotype 1 infection. Hepatol Res. 2016 Mar;46(3):E189-93. doi: 10.1111/hepr.12535. Epub 2015 Jun 18. PMID 25991083

RESULTS

PARTICIPANT FLOW:
Groups:
- 600mg Deleobuvir and 80mg Faldaprevir: Patients received 8 weeks of 600mg twice daily (bid) deleobuvir and 80 mg once daily (qd) faldaprevir (faldap) in combination with standard weight-based dose of ribavirin (RBV). Followed by 24 weeks of 120 mg once daily (qd) faldaprevir in combination with once weekly subcutaneous injection of 180 μg pegylated interferon alfa-2a (PegIFN) and standard weight-based dose of ribavirin (RBV).
- 600mg Deleobuvir and 120mg Faldaprevir: Patients received 8 weeks of 600mg twice daily (bid.) deleobuvir and 120 mg once daily (qd) faldaprevir in combination with standard weight-based dose of ribavirin (RBV). Followed by 24 weeks of 120 mg once daily (qd) faldaprevir in combination with once weekly subcutaneous injection of 180 μg pegylated interferon alfa-2a (PegIFN) and standard weight-based dose of ribavirin (RBV).
Period: Treatment Period 1: Faldap/Del/RBV
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Started | 12 | 13
Completed | 11 | 12
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Treatment Period 2: Faldap/PegIFN/RBV
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Started | 11 | 12 (One patient was treated with only PegIFN/RBV, as faldaprevir was discontinued due to adverse events)
Completed | 10 | 12
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set which included all patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Groups:
- 600mg Deleobuvir and 80mg Faldaprevir: Patients received 8 weeks of 600mg twice daily (bid) deleobuvir and 80 mg once daily (qd) faldaprevir in combination with standard weight-based dose of ribavirin (RBV). Followed by 24 weeks of 120 mg once daily (qd) faldaprevir in combination with once weekly subcutaneous injection of 180 μg pegylated interferon alfa-2a (PegIFN) and standard weight-based dose of ribavirin (RBV).
- Total: Total of all reporting groups
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir | Total
Number analyzed (Participants) | 12 | 13 | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (7.38) | 55.5 (8.42) | 56.5 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Drug-related Adverse Events
Description: Number of patients with investigator defined drug-related Adverse Events
Time Frame: From first dose of study medication until 30 days after last dose of study medication, up to 199 days
Population: as for baseline characteristics
Measure: Number; unit: participants
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 12 | 13
participants | 12 | 13

2. Secondary Outcome: Percentage of Participants With Virological Response at Week 4
Description: Percentage of participants with plasma HCV RNA (hepatitis C virus (HCV) ribonucleic acid (RNA)) level <25 IU/mL (undetected or detected) at week 4.
Time Frame: 4 weeks
Population: Full analysis set which included all patients with at least 1 on-treatment value of HCV RNA viral load
Measure: Number; unit: percentage of participants
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 12 | 13
percentage of participants | 91.7 | 92.3

3. Secondary Outcome: Percentage of Participants With Virological Response at Week 8
Description: Percentage of participants with plasma HCV RNA (hepatitis C virus ribonucleic acid ) level <25 IU/mL (undetected or detected) at week 8.
Time Frame: 8 weeks
Population: Full analysis set which included all patients with at least 1 on-treatment value of HCV RNA viral load
Measure: Number; unit: percentage of participants
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 12 | 13
percentage of participants | 91.7 | 100.0

4. Secondary Outcome: Maximum Measured Concentration (Cmax) of Deleobuvir
Description: Maximum measured concentration of BI 207127 (Deleobuvir) in plasma following the morning dose of Nth day (Cmax,N).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h, 11h 50min and 23h 50min after drug administration on days 1, 11 and 57
Population: Pharmacokinetic (PK) analysis set which included all evaluable patients. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Day 1 (N=9, 12) | 12800 (57.3) | 18800 (55.8)
  Day 11 (N=11, 12) | 30100 (71.6) | 50300 (35.4)
  Day 57 (N=11, 13) | 18800 (61.0) | 41900 (51.6)

5. Secondary Outcome: Time From Last Dosing to the Maximum Concentration (Tmax) of Deleobuvir
Description: Time from last dosing to the maximum concentration of Deleobuvir (BI 207127) in plasma after the morning dose of Nth day (Tmax,N).
Time Frame: as for outcome 4
Population: PK analysis set which included all evaluable patients. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data.
Measure: Median (Full Range); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
hours
  Day 1 (N=9, 12) | 3.97 [3.83 to 6.02] | 5.03 [1.97 to 7.87]
  Day 11 (N=11, 12) | 3.92 [1.92 to 5.92] | 3.94 [1.90 to 6.00]
  Day 57 (N=11, 13) | 4.00 [1.83 to 6.05] | 3.98 [1.97 to 6.08]

6. Secondary Outcome: Area Under the Curve (AUC) of Deleobuvir
Description: Area under the concentration time curve (AUC) of the analyte in plasma after the morning dose on the Nth day (AUCτ,N) and at steady state (AUCτ,ss), over a uniform dosing interval τ.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol*h/L
  Day 1 (N=9, 12) | 77500 (57.0) | 118000 (59.8)
  Day 11 (N=11, 12) | 216000 (104) | 404000 (52.3)
  Day 57 (N=10, 13) | 111000 (102) | 326000 (64.8)

7. Secondary Outcome: Maximum Measured Concentration (Cmax) of Faldaprevir
Description: Maximum measured concentration of Faldaprevir (BI 201335 ZW) in plasma following the morning dose of Nth day (Cmax,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
ng/mL
  Day 1 (N=9, 12) | 3380 (43.9) | 6440 (46.9)
  Day 11 (N=11, 12) | 8530 (76.0) | 20400 (39.7)
  Day 57 (N=11, 13) | 4750 (65.1) | 18700 (59.0)

8. Secondary Outcome: Time From Last Dosing to the Maximum Concentration (Tmax) of Faldaprevir
Description: Time from last dosing to the maximum concentration of Faldaprevir (BI 201335 ZW) in plasma after the morning dose of Nth day (Tmax,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
hours
  Day 1 (N=9, 12) | 3.97 [3.83 to 6.02] | 5.98 [3.97 to 23.8]
  Day 11 (N=11, 12) | 3.92 [1.92 to 9.83] | 4.00 [1.90 to 9.80]
  Day 57 (N=11, 13) | 3.92 [1.83 to 6.05] | 3.97 [1.97 to 7.93]

9. Secondary Outcome: Area Under the Curve (AUC) of Faldaprevir
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
ng*h/mL
  Day 1 (N=9, 9) | 42900 (53.0) | 107000 (36.4)
  Day 11 (N=11, 10) | 119000 (113) | 360000 (50.8)
  Day 57 (N=10, 11) | 58700 (115) | 291000 (78.5)

10. Secondary Outcome: Maximum Measured Concentration (Cmax) of BI 208333
Description: Maximum measured concentration of BI 208333 (a metabolite of Deleobuvir) in plasma following the morning dose of Nth day (Cmax,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Day 1 (N=9, 12) | 2600 (64.2) | 3630 (76.8)
  Day 11 (N=11, 12) | 11100 (92.5) | 20800 (80.5)
  Day 57 (N=11, 13) | 4630 (74.0) | 14600 (92.7)

11. Secondary Outcome: Time From Last Dosing to the Maximum Concentration (Tmax) of BI 208333
Description: Time from last dosing to the maximum concentration of BI 208333 (a metabolite of Deleobuvir) in plasma after the morning dose of Nth day (Tmax,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
hours
  Day 1 (N=9, 12) | 6.00 [3.97 to 8.00] | 7.80 [4.05 to 10.0]
  Day 11 (N=11, 12) | 5.90 [3.83 to 7.98] | 3.99 [1.83 to 8.00]
  Day 57 (N=11, 13) | 5.97 [3.87 to 6.13] | 5.98 [3.97 to 10.0]

12. Secondary Outcome: Area Under the Curve (AUC) of BI 208333
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol*h/L
  Day 1 (N=9, 12) | 19900 (67.5) | 26000 (69.5)
  Day 11 (N=11, 12) | 94200 (137) | 210000 (82.9)
  Day 57 (N=10, 13) | 38400 (109) | 141000 (112)

13. Secondary Outcome: Maximum Measured Concentration (Cmax) of CD 6168
Description: Maximum measured concentration of CD 6168 (a metabolite of Deleobuvir) in plasma following the morning dose of Nth day (Cmax,N).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h, 11h 50min and and 23h 50min after drug administration on days 1, 11 and 57
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Day 1 (N=9, 12) | 1640 (73.7) | 1920 (75.5)
  Day 11 (N=11, 12) | 12200 (144) | 23400 (40.4)
  Day 57 (N=11, 13) | 7150 (109) | 21000 (62.3)

14. Secondary Outcome: Time From Last Dosing to the Maximum Concentration (Tmax) of CD 6168
Description: Time from last dosing to the maximum concentration of CD 6168 (a metabolite of Deleobuvir) in plasma after the morning dose of Nth day (Tmax,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
hours
  Day 1 (N=9, 12) | 8.00 [6.00 to 11.9] | 9.81 [5.97 to 11.8]
  Day 11 (N=11, 12) | 3.95 [1.83 to 9.83] | 3.94 [1.90 to 6.00]
  Day 57 (N=11, 13) | 5.83 [3.85 to 6.13] | 4.10 [1.97 to 11.8]

15. Secondary Outcome: Area Under the Curve (AUC) of CD 6168
Description: as for outcome 6
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol*h/L
  Day 1 (N=8, 10) | 11200 (82.7) | 13200 (75.1)
  Day 11 (N=11, 12) | 111000 (177) | 234000 (47.5)
  Day 57 (N=10, 12) | 61400 (157) | 191000 (73.3)

16. Secondary Outcome: Maximum Measured Concentration (Cmax) of CD 6168-AG
Description: Maximum measured concentration of CD 6168-AG (a metabolite of Deleobuvir) in plasma following the morning dose of Nth day (Cmax,N). AG=acylglucuronide.
Time Frame: as for outcome 13
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Day 1 (N=9, 12) | 73.7 (81.3) | 106 (85.2)
  Day 11 (N=11, 12) | 691 (132) | 2020 (71.7)
  Day 57 (N=11, 13) | 455 (97.6) | 1780 (75.3)

17. Secondary Outcome: Time From Last Dosing to the Maximum Concentration (Tmax) of CD 6168-AG
Description: Time from last dosing to the maximum concentration of CD 6168-AG (a metabolite of Deleobuvir) in plasma after the morning dose of Nth day (Tmax,N). AG=acylglucuronide.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
hours
  Day 1 (N=9, 12) | 8.00 [7.80 to 11.8] | 9.93 [7.95 to 11.8]
  Day 11 (N=11, 12) | 5.90 [1.85 to 9.83] | 4.96 [2.00 to 9.83]
  Day 57 (N=11, 13) | 5.85 [3.85 to 6.13] | 6.08 [4.00 to 11.8]

18. Secondary Outcome: Area Under the Curve (AUC) of CD 6168-AG
Description: Area under the concentration time curve (AUC) of the analyte in plasma after the morning dose on the Nth day (AUCτ,N) and at steady state (AUCτ,ss), over a uniform dosing interval τ. AG=acylglucuronide.
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol*h/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol*h/L
  Day 1 | NA (NA) — Not calculated because parameters of 2/3rds of the subjects cannot be derived due to limitation of the data or vomiting. | NA (NA) — Not calculated because parameters of 2/3rds of the subjects cannot be derived due to limitation of the data or vomiting.
  Day 11 (N=11, 12) | 6460 (152) | 20700 (76.6)
  Day 57 (N=10, 12) | 4110 (122) | 17700 (87.2)

19. Secondary Outcome: Maximum Measured Concentration (Cmax) of RBV
Description: Maximum measured concentration of ribavirin (RBV) in plasma following the morning dose of Nth day (Cmax,N).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h and 11h 50min after drug administration on days 1 and 57
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
ng/mL
  Day 1 (N=9, 13) | 537 (27.1) | 601 (58.1)
  Day 57 (N=9, 11) | 2560 (21.8) | 2740 (31.8)

20. Secondary Outcome: Time From Last Dosing to the Maximum Concentration (Tmax) of RBV
Description: Time from last dosing to the maximum concentration of ribavirin (RBV) in plasma after the morning dose of Nth day (Tmax,N).
Time Frame: as for outcome 19
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
hours
  Day 1 (N=9, 13) | 2.00 [1.82 to 4.02] | 3.95 [1.87 to 6.05]
  Day 57 (N=9, 11) | 2.08 [1.83 to 4.13] | 2.03 [1.95 to 4.00]

21. Secondary Outcome: Area Under the Curve (AUC) of RBV
Description: Area under the concentration time curve (AUC) of ribavirin (RBV) in plasma after the morning dose on the Nth day (AUCτ,N) and at steady state (AUCτ,ss), over a uniform dosing interval τ.
Time Frame: as for outcome 19
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
ng*h/mL
  Day 1 (N=9, 13) | 3410 (19.0) | 3730 (57.6)
  Day 57 (N=8, 10) | 25700 (22.7) | 27600 (39.1)

22. Secondary Outcome: Cmax Accumulation Ratio (RA,Cmax,N) of Deleobuvir
Description: Accumulation ratio of BI 207127 (Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of Cmax after the morning dose of the Nth day and after the first dose (RA,Cmax,N), and ratio of the Cmax,ss of Deleobuvir versus itself (RA,Cmax,Met,ss).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,Cmax,11 (N=11, 12) | 2.33 (50.9) | 2.68 (47.3)
  RA,Cmax,57 (N=11, 13) | 1.46 (53.2) | 2.20 (53.6)
  RA,Cmax,Met,ss (N=11, 13) | 1.00 (0) | 1.00 (0)

23. Secondary Outcome: AUC Accumulation Ratio of Deleobuvir
Description: Accumulation ratio of BI 207127 (Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of AUC after the morning dose of the Nth day and after the first dose (RA,AUC,N), and ratio of the AUC,ss of Deleobuvir versus itself (RA,AUC,Met,ss).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,AUC,11 (N=11, 12) | 2.60 (62.5) | 3.43 (43.3)
  RA,AUC,57 (N=10, 13) | 1.21 (71.3) | 2.74 (58.9)
  RA,AUC,tau,Met,ss (N=10, 13) | 1.00 (0) | 1.00 (0)

24. Secondary Outcome: Mean Residence Time (MRTpo,ss) of Deleobuvir
Description: Mean residence time of BI 207127 (Deleobuvir) in the body after oral administration at steady state (MRTpo,ss).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h, 11h 50min and 23h 50min after drug administration on day 57
Population: Pharmacokinetic (PK) analysis set which included all evaluable patients. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data. Analysis includes patients with available data for this parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 10 | 13
hours | 6.65 (39.0) | 12.6 (52.2)

25. Secondary Outcome: Apparent Clearance (CL/F,ss) of Deleobuvir
Description: Apparent clearance of BI 207127 (Deleobuvir) in plasma following extravascular administration on the 57th day (CL/F,ss).
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litres per hour
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 10 | 13
Litres per hour | 8.25 (102) | 2.81 (64.8)

26. Secondary Outcome: Predose Measured Concentration of Deleobuvir
Description: Predose measured concentration of BI 207127 (Deleobuvir) in plasma before the morning dose of the Nth day (Cpre,N) and at steady state (Cpre,ss).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h, 11h 50min and 23h 50min after drug administration on days 11 and 57
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Cpre,11 (N=9, 12) | 10700 (217) | 23500 (61.1)
  Cpre,ss (N=11, 13) | 3280 (234) | 16599 (109)

27. Secondary Outcome: Cmax Accumulation Ratio (RA,Cmax,N) of Faldaprevir
Description: Accumulation ratio of Faldaprevir (BI 201335 ZW) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of Cmax after the morning dose of the Nth day and after the first dose (RA,Cmax,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,Cmax,11 (N=11, 12) | 2.72 (56.1) | 3.17 (55.4)
  RA,Cmax,57 (N=11, 13) | 1.51 (68.0) | 3.00 (81.7)

28. Secondary Outcome: AUC Accumulation Ratio of Faldaprevir
Description: Accumulation ratio of Faldaprevir (BI 201335 ZW) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of AUC after the morning dose of the Nth day and after the first dose (RA,AUC,N).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA, AUC,11 (N=11, 9) | 2.88 (73.0) | 3.31 (43.3)
  RA,AUC,57 (N=10, 9) | 1.28 (96.6) | 2.26 (57.6)

29. Secondary Outcome: Mean Residence Time (MRTpo,ss) of Faldaprevir
Description: Mean residence time of Faldaprevir (BI 201335 ZW) in the body after oral administration at steady state (MRTpo,ss).
  This endpoint was not analysed as the parameter was not calculable for all patients in both treatment groups.
Time Frame: as for outcome 24
Population: as for outcome 5
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 0 | 0

30. Secondary Outcome: Apparent Clearance (CL/F,ss) of Faldaprevir
Description: Apparent clearance of Faldaprevir (BI 201335 ZW) in plasma following extravascular administration on the 57th day (CL/F,ss).
Time Frame: as for outcome 24
Population: PK analysis set which included all evaluable patients. A patient was considered to be not evaluable if the patient had a protocol violation relevant to the evaluation of pharmacokinetics or had insufficient data. Analysis includes patients with available data for this parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/min
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 10 | 11
mL/min | 22.7 (114) | 6.87 (78.5)

31. Secondary Outcome: Predose Measured Concentration of Faldaprevir
Description: Predose measured concentration of Faldaprevir (BI 201335 ZW) in plasma before the morning dose of the Nth day (Cpre,N) and at steady state (Cpre,ss).
Time Frame: as for outcome 26
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
ng/mL
  Cpre,11 (N=9, 12) | 4250 (143) | 13800 (47.5)
  Cpre,ss (N=11, 12) | 1540 (176) | 9980 (92.6)

32. Secondary Outcome: Cmax Accumulation Ratio of BI 208333
Description: Accumulation ratio of BI 208333 (a metabolite of Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of Cmax after the morning dose of the Nth day and after the first dose (RA,Cmax,N), and ratio of the Cmax,ss of BI 208333 versus Cmax,ss of Deleobuvir (RA,Cmax,Met,ss).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,Cmax,11 (N=11, 12) | 3.82 (81.2) | 5.73 (36.2)
  RA,Cmax,57 (N=11, 13) | 1.60 (85.2) | 3.99 (61.2)
  RA,Cmax,Met,ss (N=11, 13) | 0.345 (24.1) | 0.349 (64.0)

33. Secondary Outcome: AUC Accumulation Ratio of BI 208333
Description: Accumulation ratio of BI 208333 (a metabolite of Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of AUC after the morning dose of the Nth day and after the first dose (RA,AUC,N), and ratio of the AUC,ss of BI 208333 versus AUC,ss of Deleobuvir (RA,AUC,Met,ss).
Time Frame: as for outcome 4
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,AUC,11 (N=11, 12) | 4.16 (106) | 8.10 (39.6)
  RA,AUC,57 (N=110 13) | 1.48 (137) | 4.92 (60.9)
  RA,AUC,tau,Met,ss (N=10, 13) | 0.345 (24.1) | 0.431 (57.9)

34. Secondary Outcome: Mean Residence Time (MRTpo,ss) of BI 208333
Description: Mean residence time of BI 208333 (a metabolite of Deleobuvir) in the body after oral administration at steady state (MRTpo,ss).
  This endpoint was not analysed as the parameter was not calculable for all patients in both treatment groups.
Time Frame: as for outcome 24
Population: as for outcome 5
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 0 | 0

35. Secondary Outcome: Predose Measured Concentration of BI 208333
Description: Predose measured concentration of BI 208333 (a metabolite of Deleobuvir) in plasma before the morning dose of the Nth day (Cpre,N) and at steady state (Cpre,ss).
Time Frame: as for outcome 26
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Cpre,11 (N=9, 13) | 7450 (186) | 16800 (87.1)
  Cpre,ss (N=11, 13) | 1630 (241) | 10700 (125)

36. Secondary Outcome: Cmax Accumulation Ratio of CD 6168
Description: Accumulation ratio of CD 6168 (a metabolite of Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of Cmax after the morning dose of the Nth day and after the first dose (RA,Cmax,N), and ratio of the Cmax,ss of CD 6168 versus Cmax,ss of Deleobuvir (RA,Cmax,Met,ss).
Time Frame: as for outcome 13
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,Cmax,11 (N=10, 12) | 8.34 (78.5) | 12.2 (71.8)
  RA,Cmax,57 (N=11, 13) | 4.90 (75.4) | 10.9 (82.5)
  RA,Cmax,Met,ss (N=11, 13) | 0.380 (47.7) | 0.500 (34.6)

37. Secondary Outcome: AUC Accumulation Ratio of CD 6168
Description: Accumulation ratio of CD 6168 (a metabolite of Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of AUC after the morning dose of the Nth day and after the first dose (RA,AUC,N), and ratio of the AUC,ss of CD 6168 versus AUC,ss of Deleobuvir (RA,AUC,Met,ss).
Time Frame: as for outcome 13
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,AUC,11 (N=10, 10) | 9.57 (74.9) | 17.0 (75.4)
  RA,AUC,57 (N=9, 11) | 5.14 (106) | 14.2 (92.5)
  RA,AUC,tau,Met,ss (N=10, 12) | 0.552 (48.0) | 0.600 (24.6)

38. Secondary Outcome: Mean Residence Time (MRTpo,ss) of CD 6168
Description: Mean residence time of CD 6168 (a metabolite of Deleobuvir) in the body after oral administration at steady state (MRTpo,ss).
  This endpoint was not analysed as the parameter was not calculable for all patients in both treatment groups.
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h, 11h 50min and and 23h 50min after drug administration on day 57
Population: as for outcome 5
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 0 | 0

39. Secondary Outcome: Predose Measured Concentration of CD 6168
Description: Predose measured concentration of CD 6168 (a metabolite of Deleobuvir) in plasma before the morning dose of the Nth day (Cpre,N) and at steady state (Cpre,ss).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h, 11h 50min and and 23h 50min after drug administration on days 11 and 57
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Cpre,11 (N=9, 13) | 9610 (246) | 17600 (76.7)
  Cpre,ss (N=11, 13) | 3190 (279) | 13100 (82.6)

40. Secondary Outcome: Cmax Accumulation Ratio of CD 6168-AG
Description: Accumulation ratio of CD 6168-AG (a metabolite of Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of Cmax after the morning dose of the Nth day and after the first dose (RA,Cmax,N), and ratio of the Cmax,ss of CD 6168-AG versus Cmax,ss of Deleobuvir (RA,Cmax,Met,ss). AG=acylglucuronide.
Time Frame: as for outcome 13
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,Cmax,11 (N=11, 8) | 10.8 (105) | NA (NA) — Not calculable as per Boehringer Ingelheim internal rules summary statistics are not calculated when less than 2/3rds of patients have available data.
  RA,Cmax,57 (N=11, 13) | 7.11 (109) | 17.2 (89.8)
  RA,Cmax,Met,ss (N=11, 13) | 0.0242 (45.4) | 0.0424 (53.9)

41. Secondary Outcome: AUC Accumulation Ratio of CD 6168-AG
Description: Accumulation ratio of CD 6168-AG (a metabolite of Deleobuvir) in plasma after the administration of the Nth day over a uniform dosing interval tau, expressed as a ratio of AUC after the morning dose of the Nth day and after the first dose (RA,AUC,N), and ratio of the AUC,ss of CD 6168-AG versus AUC,ss of Deleobuvir (RA,AUC,Met,ss). AG=acylglucuronide.
Time Frame: as for outcome 13
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
Ratio
  RA,AUC,11 (N=11, 8) | 16.7 (122) | NA (NA) — Not calculable as per Boehringer Ingelheim internal rules summary statistics are not calculated when less than 2/3rds of patients have available data.
  RA,AUC,57 (N=9, 8) | 8.06 (163) | NA (NA) — Not calculable as per Boehringer Ingelheim internal rules summary statistics are not calculated when less than 2/3rds of patients have available data.
  RA,AUC,tau,Met,ss (N=10, 12) | 0.0369 (36.6) | 0.0557 (46.2)

42. Secondary Outcome: Mean Residence Time (MRTpo,ss) of CD 6168-AG
Description: Mean residence time of CD 6168-AG (a metabolite of Deleobuvir) in the body after oral administration at steady state (MRTpo,ss). AG=acylglucuronide.
  This endpoint was not analysed as the parameter was not calculable for all patients in both treatment groups.
Time Frame: as for outcome 38
Population: as for outcome 5
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 0 | 0

43. Secondary Outcome: Predose Measured Concentration of CD 6168-AG
Description: Predose measured concentration of CD 6168-AG (a metabolite of Deleobuvir) in plasma before the morning dose of the Nth day (Cpre,N) and at steady state (Cpre,ss). AG=acylglucuronide.
Time Frame: as for outcome 39
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nmol/L
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
nmol/L
  Cpre,11 (N=9, 13) | 566 (154) | 1630 (73.9)
  Cpre,ss (N=11, 13) | 211 (197) | 1350 (82.8)

44. Secondary Outcome: AUC Accumulation Ratio of RBV
Description: Accumulation ratio of ribavirin (RBV) in plasma after the administration of the 57th day over a uniform dosing interval tau, expressed as a ratio of AUC after the morning dose of the 57th day and after the first dose (RA,AUC,57).
Time Frame: as for outcome 19
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 8 | 10
Ratio | 8.03 (17.5) | 6.89 (60.8)

45. Secondary Outcome: Cmax Accumulation Ratio (RA,Cmax,57) of RBV
Description: Accumulation ratio of ribavirin (RBV) in plasma after the administration of the 57th day over a uniform dosing interval tau, expressed as a ratio of Cmax after the morning dose of the 57th day and after the first dose (RA,Cmax,57).
Time Frame: as for outcome 19
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 9 | 11
Ratio | 5.05 (22.5) | 4.89 (67.6)

46. Secondary Outcome: Mean Residence Time (MRTpo,ss) of RBV
Description: Mean residence time of ribavirin (RBV) in the body after oral administration at steady state (MRTpo,ss).
  This endpoint was not analysed as the parameter was not calculable for all patients in both treatment groups.
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h and 11h 50min after drug administration on day 57
Population: as for outcome 5
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 0 | 0

47. Secondary Outcome: Predose Measured Concentration of RBV
Description: Predose measured concentration of ribavirin (RBV) in plasma before the morning dose of the Nth day (Cpre,N) and at steady state (Cpre,ss).
Time Frame: 10 minutes (min) before drug administration and 2 hours (h), 4h, 6h, 8h, 10h and 11h 50min after drug administration on days 11 and 57
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | 600mg Deleobuvir and 80mg Faldaprevir | 600mg Deleobuvir and 120mg Faldaprevir
Number analyzed (Participants) | 11 | 13
ng/mL
  Cpre,11 (N=9, 13) | 1400 (26.8) | 1290 (31.8)
  Cpre,ss (N=10, 12) | 2080 (25.6) | 2110 (38.6)

ADVERSE EVENTS:
Time Frame: From first dose of study medication until 30 days after last dose of study medication, up to 199 days
Groups:
- Faldap/Del/RBV:80mg Faldap and 600mg Del.: Patients received 8 weeks of 600mg twice daily (bid) deleobuvir (del) and 80 mg once daily (qd) faldaprevir (faldap) in combination with standard weight-based dose of ribavirin (RBV)
- Faldap/Del/RBV:120mg Faldap and 600mg Del.: Patients received 8 weeks of 600mg twice daily (bid.) deleobuvir (del) and 120 mg once daily (qd) faldaprevir (faldap) in combination with standard weight-based dose of ribavirin (RBV)
- Faldap/pegIFN/RBV:80mg Faldap and 600mg Del.: Patients received 24 weeks 120 mg once daily (qd) faldaprevir (faldap) in combination with once weekly subcutaneous injection of 180 μg pegylated interferon alfa-2a (PegIFN) and standard weight-based dose of ribavirin (RBV), following treatment of 8 weeks of 600mg twice daily (bid) deleobuvir (del) and 80 mg once daily (qd) faldaprevir (faldap) in combination with standard weight-based dose of ribavirin (RBV).
- Faldap/pegIFN/RBV:120mg Faldap and 600mg Del.: Patients received 24 weeks 120 mg once daily (qd) faldaprevir in combination with once weekly subcutaneous injection of 180 μg pegylated interferon alfa-2a (PegIFN) and standard weight-based dose of ribavirin (RBV), following treatment of 8 weeks of 600mg twice daily (bid.) deleobuvir (del) and 120 mg once daily (qd) faldaprevir (faldap) in combination with standard weight-based dose of ribavirin (RBV).
Arm/Group | Faldap/Del/RBV:80mg Faldap and 600mg Del. | Faldap/Del/RBV:120mg Faldap and 600mg Del. | Faldap/pegIFN/RBV:80mg Faldap and 600mg Del. | Faldap/pegIFN/RBV:120mg Faldap and 600mg Del.
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 1/11 | 0/12
Other Adverse Events (participants affected / at risk) | 12/12 | 13/13 | 11/11 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Faldap/Del/RBV:80mg Faldap and 600mg Del. (N=12) | Faldap/Del/RBV:120mg Faldap and 600mg Del. (N=13) | Faldap/pegIFN/RBV:80mg Faldap and 600mg Del. (N=11) | Faldap/pegIFN/RBV:120mg Faldap and 600mg Del. (N=12)
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Faldap/Del/RBV:80mg Faldap and 600mg Del. (N=12) | Faldap/Del/RBV:120mg Faldap and 600mg Del. (N=13) | Faldap/pegIFN/RBV:80mg Faldap and 600mg Del. (N=11) | Faldap/pegIFN/RBV:120mg Faldap and 600mg Del. (N=12)
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 0 | 1 | 1 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 1
Retinal tear (Eye disorders) | 0 | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 0 | 2 | 0
Scintillating scotoma (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 4 | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 10 | 3 | 1
Oral discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Vomiting (Gastrointestinal disorders) | 4 | 8 | 2 | 2
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1
Injection site erythema (General disorders) | 1 | 0 | 0 | 0
Injection site pain (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 0 | 0 | 0 | 3
Malaise (General disorders) | 2 | 0 | 2 | 1
Mass (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 3
Pyrexia (General disorders) | 0 | 1 | 2 | 3
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 4 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 2 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 2 | 3 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 3 | 2
Red blood cell count decreased (Investigations) | 0 | 1 | 2 | 0
Weight decreased (Investigations) | 0 | 2 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 5 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 3 | 2
Hypoaesthesia (Nervous system disorders) | 2 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Depressive symptom (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photodermatosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 3 | 4 | 2
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 7 | 3 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Tanning (Social circumstances) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.